CLINICAL TRIAL: NCT05339490
Title: Evaluation of the Safety and Effectiveness of Progenitor Biological Bandages in Burn Care
Brief Title: Use of Progenitor Biological Bandages in Burn Care (Bru_PBB)
Acronym: Bru_PBB
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Following issues with the quality of the clinical cell banks used to manufacture the biological dressings, we decided not to implement this research to not compromise neither the patient safety, nor the expected efficacy of the treatment.
Sponsor: Dr Anthony De Buys Roessingh (Other)
Responsible Party: Sponsor-Investigator, Dr Anthony De Buys Roessingh, Principal investigator, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RA10106; 2020-01873 (Other: Cantonal Commission (Vaud) on Ethics in Human Research); 2020TpP1010 (Other: Swiss Agency for Therapeutic Products)
Record Dates: First submitted 2022-04-04; First posted 2022-04-21 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Burn Injury
Keywords: cell therapies; fetal progenitor cells; regenerative medicine; standardized transplants; wound healing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Progenitor Biological Bandages (Experimental): Donor Site Wound (DSW) is created with a dermatome. PBB are placed on the wound and maintained in place with the help of classical bandages for a maximum of 15 ± 1 days.
  Dressing's changes are performed at Day 5 ± 1 and Day 10 ± 1.
  Interventions: Drug: Progenitor Biological Bandages
- Jelonet (Active Comparator): Donor Site Wound is created with a dermatome. Jelonet® are placed on the wound and maintained in place with the help of classical bandages for a maximum of 15 ± 1 days.
  Dressing's changes are performed at Day 5 ± 1 and Day 10 ± 1.
  Interventions: Device: Jelonet

INTERVENTIONS:
Drug: Progenitor Biological Bandages — The patients candidates for a skin autograft and a consequent Donor Site Wound (DSW) creation with a dermatome will be randomized between 2 treatment arms. As soon as DSW is created and according to randomization results, PBB will be placed on the wound and maintained in place with the help of classical bandages for a maximum of 15 ± 1 days with dressing's changes at Day 5 ± 1 and Day 10 ± 1. Old PBB will be replaced by new ones according to the local procedure.
  Pictures will be taken at each change and on-site evaluation of the wound healing (% of re-epithelialization) will be done by the surgeon. If the DSW is not closed at D15 ± 1, Jelonet® will be used to cover the skin until complete skin closure. If the wound is closed after 15 ± 1 days or before, the scar will then be topically treated with cream as standard treatment. All patients will be followed until 5 years according to the long-term evaluation calendar to monitor long-term skin quality.
  Other Names: PBB
  Arms: Progenitor Biological Bandages
Device: Jelonet — The patients candidates for a skin autograft and a consequent Donor Site Wound (DSW) creation with a dermatome will be randomized between 2 treatment arms. As soon as DSW is created and according to randomization results, Jelonet, as standard bandages, will be placed on the wound and maintained in place with the help of classical bandages for a maximum of 15 ± 1 days with dressing's changes at Day 5 ± 1 and Day 10 ± 1.
  Pictures will be taken at each change and on-site evaluation of the wound healing (% of re-epithelialization) will be done by the surgeon. If the DSW is not closed at D15 ± 1, Jelonet® will be used to cover the skin until complete skin closure. If the wound is closed after 15 ± 1 days or before, the scar will then be topically treated with cream as standard treatment. All patients will be followed until 5 years according to the long-term evaluation calendar to monitor long-term skin quality.
  Arms: Jelonet

SUMMARY:
Skin, as the outermost organ of the human body, serves as a protective layer from microorganisms and external forces, and allows controlling fluid loss among other important functions (sensory, immune and aesthetic functions). When the skin is burned, the extent of the depth can be classified in 1rst, 2nd superficial to deep, 3rd and 4th degree burns, according to the different layers of the skin and tissue that are affected in depth. Severity of a burn can also be characterized by total body surface area (TBSA), location of the burn injury, subject characteristics and age according to the European Practice Guidelines for Burn Care. The actual gold standard treatment for 3rd or deep 2nd degree burn wounds is skin autografting that means transplantation of healthy skin taken from an undamaged donor site on the patient to the wound site, therefore creating a donor site wound (DSW).

The Burn Center of the CHUV has developed Progenitor Biological Bandages (PBB), composed of human skin progenitor cells (produced and stored GMP clinical cell bank with the Hospital accredited Cell Production Center, CPC) seeded on a biodegradable collagen scaffold (Resorba®), to support wound healing of DSW, as well as 2nd degree burn wounds. PBB have been applied at the CHUV under emergency circumstances over the last 20 years in children and adults with a TBSA higher than 10% and 20%, respectively.

These PBB aim to increase the spontaneous healing of 2nd superficial and deep burns to avoid the skin autograft, and therefore prevent the creation of a second wound with the DSW. Furthermore, if skin grafting cannot be avoided, in the case of a 3rd or 2nd degree deep burns that do not close spontaneously, the use of PBB is an advantage for treating DSW in order to accelerate its healing process and therefore use the same donor site for future treatments.

The aim of this study is to demonstrate the efficacy of the PBB treatment of the DSW compared to standard-care treatment (Jelonet®), and therefore verify our hypothesis of higher performance of PBB. The investigators would like also to assess the efficacy of the DSW treatment on short- and long-term periods, as well as to collect observational data on 2nd degree burn wound treated with PBB. Furthermore, another objective of this study is to confirm the safety of the PBB on DSW and 2nd degree burn wounds.

DETAILED DESCRIPTION:
Study Product / Intervention:

PBB (Progenitor Biological Bandages) produced at CHUV by the Cell Production Center are single-use therapies, which are applied on 2nd degree burns, defined as superficial to partial-thickness burns, and DSW (Donor Site Wound). They can be applied on complex anatomies (moldable) in adults and children of both genders after cleaning of the wounds through showering and debridement. The application of these PBB is prescribed by a specialized surgeon to a patient incapable of spontaneous burn closure and they are only used by health professionals at the CHUV Burn Center. PBB are composed of human skin progenitor cells (FE002- SK2 cell type) originated from a clinical GMP cell bank and seeded on a biodegradable horse collagen scaffold (9x12 cm, Resorba® Medical). PBB are delivered directly to the surgeon in the operating room after a production period of at least 18 hours. The number of PBB ordered by the physician depends on the burned surface area to be treated. They are maintained in the appropriate medium in controlled conditions until delivery and application. They must be applied no later than 72 hours after the start of production. Treatment duration with PBB is 10-12 days post injury for 2nd degree burn wounds and 15 days post DSW creation for DSW.

Control Intervention (if applicable):

To evaluate the performance of treatment with PBB, the investigators plan to compare in a randomization process the efficacy of PBB against a control intervention with Jelonet®. Jelonet® is the standard treatment for treating a DSW when a skin autograft is needed for 2nd and 3rd degree burned patients. The DSW is performed by using a dermatome (Aesculap®, Braun) to retrieve healthy skin (0.2 mm depth) when a skin graft is required to treat burn wound. The DSW is similar to a 2nd degree superficial burn and is able to heal by treatment with Jelonet® dressings (Paraffin Gauze Dressings, 10cm x 10 cm, Smith & Nephew, UK). The advantage to compare treatments efficacies on a DSW is due to the homogenous properties of a DSW, in comparison to the heterogeneous aspect of a burn wound. Treatment duration of DSW with Jelonet® is 15 days after the creation of DSW.

Measurements and procedures:

Interventional/Comparative cohort (adult and pediatric patients with 2nd or 3rd degree burns treated with a skin autograft):

* Treatment group "Donor site wound": treatment with PBB
* Control group "Donor site wound": treatment with Jelonet® The participants who will be candidates for a skin autograft and a consequent DSW creation with a dermatome will be randomized for the treatment of DSW between PBB and Jelonet® in order to verify the hypothesis of higher performance of PBB in the skin healing process. As soon as the DSW is created, PBB or Jelonet® will be placed on the wound and maintained in place with the help of classical bandages for a maximum of 15 ± 1 days with dressing's changes at Day 5 ± 1 and Day 10 ± 1. In case of the use of PBB, old bandages will be replaced by new ones according to the procedure. When Jelonet® is used, it may occur that the bandage remains adherent to un-epithelialized area. In that case, the edges of the Jelonet® that have peeled off (i.e. where the wound has re-epithelialized) will be cut and new bandages will be applied. Pictures will be taken at each change and on-site evaluation of the wound healing (% of re-epithelialization) will be done by the investigators. If the DSW is not closed at D15 ± 1, Jelonet® will be used to cover the skin until complete skin closure. If the wound is closed after 15 ± 1 days or before, the scar will then be topically treated with cream as standard treatment. All participants will be followed until 5 years according to the long-term evaluation calendar to monitor long-term skin quality.

Interventional/Observational cohort (adult and pediatric patients with 2nd degree burns treated with PBB):

• Treatment group "Burn wound": treatment with PBB For the participants with 2nd degree burns, a first-line treatment of the wounds with PBB as first cover will be prescribed by the surgeon during the first 10- 12 days post injury with maximum 4 dressings' changes every 2-3 days. Old bandages will be replaced by new ones according to the procedure. Pictures will be taken at each bandage change and on-site evaluation of the wound healing will be done by the investigators (% of re-epithelialization). If after 10-12 days, the wound is not closed (95% re-epithelialization not achieved), then the surgeon will decide to perform a skin autograft to help the healing process. If the wound is closed after 10-12 days or before, the scar will then be topically treated with cream. In the case a 2nd degree burn treated with PBB progresses to a 3rd degree burn, the treatment options will be discussed again during treatment and a skin autograft will be performed. All participants will be followed until 5 years post injury according to the long-term evaluation calendar to monitor long-term skin quality.

ELIGIBILITY:
Inclusion Criteria:

* ≤ 2 years old with ≥5% TBSA
* between 3 and 10 years old with ≥10% TBSA
* between 11 and 18 years old with ≥15% TBSA
* ≥ 18 years old with ≥ 20% TBSA
* ≥ 65 years old with ≥ 10% TBSA
* Any age with burns on the face, hands, genitalia or major joints
* Patient with 2nd (superficial to deep) degree burn wounds
* Patient with 3rd degree burns candidate for a skin autograft
* Informed Consent as documented by signature and according to consent in case of emergency situation
* First injury
* Possibility of Follow-up for 5 years after injury

Exclusion Criteria:

* Infected wounds
* Vitally unstable patients
* Known allergy or hypersensitivity to product of equine origin
* Refusal of the study by the participants or relatives

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Wound re-epithelialization assessment at Day 10 | Day 10 of treatment
  95 percent skin re-epithelialization (yes or no) will be assessed 10 days after the start of treatment and creation of the DSW

SECONDARY OUTCOMES:
Short-term efficacy of treatment | Day 5, Day 10, and Day 15 of treatment
  Percentage of re-epithelialization (percent) by measuring the length (cm) and height (cm) of the wound at each evaluation time point compared to Day 1 of treatment
Long-term skin quality - Scar appearance (Vancouver Scar Scale) | From 1 month to 5 years post skin closure
  The Vancouver scale allows to measure scar appearance by evaluation of scores for:
  * skin pliability (0=Normal; 1=Supple; 2=Yielding; 3=Firm; 4=Adherent),
  * skin vascularization (0=Normal; 1=Pink; 2=Red; 3=Purple)
  * skin pigmentation (0=Normal; 1=Hypopigmentation; 2=Mixed; 3=Hyperpigmentation). The quality of the skin is assessed both by vision and touch by medical experts for a better standardization. Higher scores mean a worse outcome.
Long-term skin quality - Scar colour | From 1 month to 5 years post skin closure
  Scar colour will be evaluated with a probe-based skin analysis system from Cortex Technology. The erythema and melanin indexes (EI and MI) are read directly on the device with arbitrary units specific to the device (between 0 and 100).
Long-term skin quality - Elastography | From 1 month to 5 years post skin closure
  Elastic properties of the repaired skin (m/s) using a probe-based skin analysis system from Cortex Technology will be measured and compared to healthy skin.

OTHER OUTCOMES:
Safety outcomes - wound infections | Through study treatment, an average of 15 days for each treated wounds
  Incidence of wound infections will be monitored according to microbiological assessment on tissue biopsy in case of infection suspicion of the wound.
Safety outcomes - adverse events | Through study completion, an average of 5 years
  Incidence of adverse events from initial treatment through last study visit. The AEs and SAEs will be assessed by the physician (type, duration, severity, relationship to the investigational medicinal product and need for treatment) and graded according to the CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Anthony De Buys Roessingh, Principal Investigator — Lausanne Burn Center, Lausanne University Hospital CHUV
Locations (1):
- University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hohlfeld J, de Buys Roessingh A, Hirt-Burri N, Chaubert P, Gerber S, Scaletta C, Hohlfeld P, Applegate LA. Tissue engineered fetal skin constructs for paediatric burns. Lancet. 2005 Sep 3-9;366(9488):840-2. doi: 10.1016/S0140-6736(05)67107-3. PMID 16139659
- [Background] De Buys Roessingh AS, Hohlfeld J, Scaletta C, Hirt-Burri N, Gerber S, Hohlfeld P, Gebbers JO, Applegate LA. Development, characterization, and use of a fetal skin cell bank for tissue engineering in wound healing. Cell Transplant. 2006;15(8-9):823-34. doi: 10.3727/000000006783981459. PMID 17269452
- [Background] Abdel-Sayed P, Michetti M, Scaletta C, Flahaut M, Hirt-Burri N, de Buys Roessingh A, Raffoul W, Applegate LA. Cell therapies for skin regeneration: an overview of 40 years of experience in burn units. Swiss Med Wkly. 2019 May 19;149:w20079. doi: 10.4414/smw.2019.20079. eCollection 2019 May 6. PMID 31104308
- [Background] Abdel-Sayed P, Hirt-Burri N, de Buys Roessingh A, Raffoul W, Applegate LA. Evolution of Biological Bandages as First Cover for Burn Patients. Adv Wound Care (New Rochelle). 2019 Nov 1;8(11):555-564. doi: 10.1089/wound.2019.1037. Epub 2019 Oct 16. PMID 31637102
- [Background] Laurent A, Lin P, Scaletta C, Hirt-Burri N, Michetti M, de Buys Roessingh AS, Raffoul W, She BR, Applegate LA. Bringing Safe and Standardized Cell Therapies to Industrialized Processing for Burns and Wounds. Front Bioeng Biotechnol. 2020 Jun 19;8:581. doi: 10.3389/fbioe.2020.00581. eCollection 2020. PMID 32637400